CLINICAL TRIAL: NCT01941537
Title: A Randomized Placebo-controlled Study to Determine the Safety, Tolerability, Pharmacodynamics and Clinical Efficacy of ILV-094 (an IL-22 Antibody) Administered Intravenously to Subjects With Atopic Dermatitis (AD)
Brief Title: Randomized Placebo Controlled Study to Determine Safety, Pharmacodynamics and Efficacy of ILV-094 in Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JKR-0766
Record Dates: First submitted 2013-08-29; First posted 2013-09-13 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-01

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — fezakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ILV-094 (Experimental): Forty patients will be enrolled in the ILV-094 treatment arm. A loading IV dose of 600 mg of ILV-094 will be given at baseline (Day 0), followed by five additional IV doses of 300 mg of ILV-094 every two weeks (Weeks 2, 4, 6, 8, and 10).
  Interventions: Drug: ILV-094
- Placebo comparator (Placebo Comparator): Twenty patients will be enrolled in the ILV-094 placebo arm. A loading IV dose of placebo will be given at baseline (Day 0), followed by five additional IV doses of placebo every two weeks (Weeks 2, 4, 6, 8, and 10).
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: ILV-094 — IV infusion of ILV-094
  Arms: ILV-094
Drug: Placebo Comparator — Twenty patients will be enrolled in the ILV-094 placebo arm. A loading IV dose of a placebo will be given at baseline (Day 0), followed by five additional IV doses of placebo every two weeks (Weeks 2, 4, 6, 8, and 10).
  Other Names: Placebo
  Arms: Placebo comparator

SUMMARY:
Atopic dermatitis (AD) is a common inflammatory skin disorder that adversely affects most aspects of everyday life in majority of patients. It has a prevalence of up to 3-4% of adults and up to 25% among children. AD has a complex pathogenesis, characterized by: 1) immune activation with increased numbers of T-cells, dendritic cells (DCs), and increased expression of inflammatory molecules 2) marked epidermal hyperplasia in chronic diseased skin, and 3) defective barrier function with increased trans-epidermal water loss (TEWL) and decreased lipids, reflecting underlying alterations in keratinocyte differentiation. AD is predominantly a Th2 (IL-4, IL-13, and IL-31) disease, and recently was also found to be a "T22" (IL-22) polarized disease.

ILV-094 is an anti IL-22 antibody and therefore should reverse the immune activation of AD. This study is being done to assess the safety, tolerability, clinical efficacy, and mechanism of action of ILV-094 in patients with AD.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, study of six IV infusions of ILV-094 administered to subjects with atopic dermatitis. Sixty subjects will be randomly assigned in a 2:1 ratio to one of the two treatments arms (ILV-094 vs placebo). Forty patients will be enrolled in the ILV-094 treatment arm and 20 in the placebo-treatment arm, accordingly. A loading IV dose of 600 mg of ILV-094 or placebo will be given at baseline (Day 0), followed by five additional IV doses of 300 mg of ILV-094 or placebo every two weeks (Weeks 2, 4, 6, 8, and 10). We will continue to follow the patients every two weeks for an additional 10 weeks after the last IV dose (20 weeks post baseline).

ELIGIBILITY:
-Inclusion Criteria:

Signed and dated an IRB-approved informed consent form before any study-specific screening procedures are performed.

Male or females between the ages of 18-75 year-old.

Have moderate to severe AD (as determined using the Objective SCORAD scale ≥30), and an IGA index>3).

Patients who fail or cannot sustain response with one or more of the three treatment categories listed below (used for at least 4 weeks):

* Category 1: Hydration plus topical steroids and/or antibiotics (tetracycline, bactrim, cephalosporins, etc) and or topical immune modulators (protopic/elidel).
* Category 2: Systemic Steroids and/or Phototherapy.
* Category 3: Cyclosporine and/or Other Immunomodulators (Methotrexate, CellCept, and Immuran).
* A washout period from cyclosporine and/or oral steroids of 4 weeks and from phototherapy of 2 weeks prior to baseline.
* A washout period of at least 1 week prior to baseline will also be required for patients that responded, but did not sustain response to strong topical steroids (i.e clobetasol) or topical immune modulators (i.e Protopic, and Elidel).
* The patients will be allowed to use topical therapy during the washout period. These will include emollients, and mild steroids (class 6 or 7), except on one target area that will be the site for the skin biopsies.
* A washout period from any systemic investigational therapy of at least 90 days.
* A washout period from cyclosporine and/or oral steroids of 4 weeks and from phototherapy of 2 weeks prior to baseline.
* A washout period of at least 1 week prior to baseline will also be required for patients that responded, but did not sustain response to strong topical steroids (i.e clobetasol) or topical immune modulators (i.e protopic, and elidel).
* The patients will be allowed to use topical therapy during the washout period. These will include emollients, and mild steroids (class 6 or 7), except on one target area that will be the site for the skin biopsies.

Women of childbearing potential must test negative for pregnancy and agree to use birth control measures that are highly effective. Highly effective methods are defined as those that result in a low failure rate (i.e. less that 1 percent per year abstinence) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices (IUD's), sexual abstinence, or a vasectomized partner. Likewise, sexually active men must also use appropriate methods of birth control (e.g., abstinence, barrier methods with spermicide, or have had surgical sterilization such as vasectomy).

PPD negative at screening.

Patients with stable chronic asthma, treated with inhaled corticosteroids, will be allowed to participate in the study.

Willingness to avoid alcohol intake 48 hours before each visit in which study drug will be received, in order to avoid increases in liver function tests (LFTs) (this was an exclusion in other ILV-094 studies in order to guard against increased LFTs due to alcohol intake being attributed to study drug).

-Exclusion Criteria:

History of active or latent serious infections (TB, or other granulomatous disorders such as histoplasmosis, coccidioidomycosis, etc). Skin colonization by Staph. aureus is expected in a high percentage of atopic patients with active disease and will not be considered as an exclusion criteria.

*Patients with a history of a positive PPD that have received prophylaxis will be permitted to enroll into the study.

Have a known malignancy or history of malignancy (except for basal or squamous cell carcinoma completely excised without evidence of recurrence and treated carcinoma in situ of the cervix) or lymphoproliferative diseases such as including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (e.g. nodes in the posterior triangle of the neck, intraclavicular, epitrochlear or periaortic areas) or splenomegaly.

Have a nontuberculous mycobacterial infection or opportunistic systemic infection (e.g., Pneumocystis carinii, and aspergillosis) within 6 months prior to screening.

Have positive HIV by history or POCT on the screening visit.

Have documented current active hepatitis B (surface antigen positive or asymptomatic chronic carriers) or a history of hepatitis C infection (anti-HCV positive), by history and/or screening test.

Have a history of substance abuse (drug or alcohol) within the past year before screening.

Have a serious concomitant illness that could require the use of systemic corticosteroids or otherwise interfere with the patient's participation in the trial.

Pregnant women or women that are breast feeding or plan to breast feed.

Evidence of acute or unstable clinically significant disease (eg, unstable cardiovascular, cerebrovascular, respiratory, renal, or psychiatric disease or any unstable serious disorder requiring active frequent monitoring.

Evidence of other concomitant skin conditions (eg, psoriasis, or lupus erythematosus) other than atopic dermatitis that would interfere with evaluations of the effect of study medication on atopic dermatitis.

Have shown a previous immediate hypersensitivity response, including anaphylaxis, to an immunoglobulin product (plasma-derived, recombinant, e.g. monoclonal antibody).

Use of any investigational small molecule drug within 90 days before the first dose of test article administration.

Have a transplanted organ (with the exception of a corneal transplant performed >3 months prior to screening).

Have concomitant autoimmune disease (such as lupus, rheumatoid arthritis, multiple sclerosis, Crohn's Disease, etc).

Clinically important deviation from normal limits in physical examination, vital sign measurements, 12-lead electrocardiograms (ECGs), or clinical laboratory tests results, not associated with a chronic, well-controlled medical condition. Examples of these

deviations include following:

1. Undiagnosed hypertension.
2. Evidence of undiagnosed ischemic heart disease or potentially

   clinically significant arrhythmia on ECG.
3. Hemoglobin <9 g/dl
4. WBC count < 3.5 x 109 cells/L
5. Neutrophils <1 x 109 cells/L
6. Platelets < 100 x 109 cells/L
7. AST/SGOT and ALT/SGPT levels above 2 times the upper limit of normal for the laboratory conducting the test.
8. Alkaline phosphatase levels above 2 times the upper limit of normal for the laboratory conducting the test.

Live vaccines within 3 months before test article administration or during the study.

Any medical, psychological or social condition that, in the opinion of the investigator, would jeopardize the health or well-being of the participant during any study procedures or the integrity of the data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Krueger, MD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ILV-094 | Placebo Comparator
Started | 40 | 20
Completed | 36 | 17
Not Completed | 4 | 3
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ILV-094 | Placebo Comparator | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 20 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (14.9) | 41.3 (16.3) | 40.5 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 23 | 9 | 32
Region of Enrollment [Number; unit: participants]
  United States | 40 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in SCORAD
Description: Percentage Change in the Scoring of Atopic Dermatitis (SCORAD) at week 12 compared to baseline in both arms of the study in subjects with atopic dermatitis.
  SCORAD (Severity scoring of Atopic Dermatitis) is composite severity index comprising a) the amount/extent of body surface area affected, b) subjective symptom visual analog assessments [itchy 0 (no itching) to 3 (severe itching) and sleep disturbance 0(no sleep disturbance) to 3 (severe sleep disturbance)], and c) 6 disease intensity assessments [dryness/scaling, erythema, induration/papulation, excoriation, lichenification and oozing/weeping/crusting, each graded from 0 to (none) to 3 (severe). A SCORAD score ranges from 0 (no AD present) to 103 (severe).
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | ILV-094 | Placebo Comparator
Number analyzed (Participants) | 40 | 20
percentage change | -18.8 (2.9) | -11.7 (3.9)

2. Secondary Outcome: The Percentage of Patients Who Achieve an Improvement of 50% or Greater From Their Baseline Objective SCORAD at Week 12 of ILV-094 Treatment
Description: The SCORAD50 captures individuals who achieved 50% or greater improvement from baseline SCORAD score. This outcome measure is the percentage of participants who achieved SCORAD50 at week 12. This analysis will be performed using fisher exact test. Patients who drop-out will be considered treatment failures (non-responder approach). A sensitivity analysis will be carried out using data as observed.
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | ILV-094 | Placebo Comparator
Number analyzed (Participants) | 40 | 20
percentage of participants | 22.2 | 15.0

3. Secondary Outcome: The (Per-patient) Percent Improvement in the SCORAD Relative to Baseline.
Description: The (per-patient) percent improvement in the SCORAD relative to baseline, which will be analyzed using the MMRM approach described for the primary efficacy endpoint. Improvement is measured as the reduction in the score.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: percentage decline in SCORAD score
Arm/Group | ILV-094 | Placebo Comparator
Number analyzed (Participants) | 40 | 20
percentage decline in SCORAD score | -13.8 (2.7) | -8.0 (3.1)

4. Secondary Outcome: Change in IGA Score
Description: Change in Investigator Global Assessment score (IGA) at week 12 as compared to baseline for both arms of the study in subjects with atopic dermatitis.
  IGA is a score between 0-5, with 0 being all clear, 1 being almost clear, 2 being mild disease, 3 being moderate disease, 4 being severe disease and 5 being very severe disease.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ILV-094 | Placebo Comparator
Number analyzed (Participants) | 40 | 20
score on a scale | -0.6 (0.1) | -0.3 (0.1)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | ILV-094 | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 2/40 | 0/20
Other Adverse Events (participants affected / at risk) | 4/40 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ILV-094 (N=40) | Placebo Comparator (N=20)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) — Pregnancy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ILV-094 (N=40) | Placebo Comparator (N=20)
Mild Adverse Event (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) — Upper respiratory infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes